CLINICAL TRIAL: NCT03603015
Title: Contractility: Cuff Versus Urodynamics Testing In Males With Voiding Lower Urinary Tract Symptoms
Acronym: CONCUR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Newcastle-upon-Tyne Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 8598
Record Dates: First submitted 2018-06-27; First posted 2018-07-27 (Actual); Last update posted 2018-09-17 (Actual); Status verified 2018-09

CONDITIONS: Lower Urinary Tract Symptoms
Keywords: bladder; urinary tract; symptoms; contractility; urodynamics; penile cuff test
MeSH Terms: conditions — Lower Urinary Tract Symptoms

STUDY DESIGN:
Intervention Model Description: Single pilot group all receiving the same tests
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pilot group: urodynamics and cuff test (Other): Single-arm study with all participants undergoing cystometrogram, then cystometrogram with simultaneous penile cuff test, then penile cuff test alone
  Interventions: Diagnostic Test: Penile cuff test

INTERVENTIONS:
Diagnostic Test: Penile cuff test — Comparison of invasive vs non-invasive urodynamics
  Other Names: Cystometrogram

SUMMARY:
A number of men will experience bothersome urinary symptoms, which become more common as they age. A number of conditions can cause these symptoms, and general practitioners may refer men to their local hospital for further assessment and treatment. Symptoms can include poor flow of urine, the need to pass urine more frequently, or the sensation that the bladder is not completely emptying. This can be due to an enlargement of the prostate gland. These symptoms can also be caused when the bladder muscle is not able to contract (squeeze) as well as it previously has to empty the bladder. This is known as underactive bladder (UAB).

It is important to distinguish between the two conditions as a cause for these symptoms, to prevent side effects from unnecessary medications or operations. Currently, men would need to undergo a bladder pressure test (urodynamics). This involves inserting a catheter via the penis into the bladder, through which the bladder is filled with fluid and pressure is measured. A separate second small tube is inserted into the rectum to measure the pressure in the abdomen. The pressure changes are observed as the bladder is filled, and then urine is passed around the catheter.

A second technique for measuring bladder pressure is the use of a small inflatable cuff which is placed around the penis (penile cuff test). The bladder pressure can then be determined by inflating the cuff and interrupting the flow of urine. The bladder can be filled naturally before the test, which means a bladder catheter tube is not required. This study is designed to find out ways that the penile cuff test can be made more accurate. It will compare the cuff results to those obtained from a bladder pressure test, and will take x-ray pictures of the urinary tract during the test.

DETAILED DESCRIPTION:
The investigators intend to refine the procedural steps of the cuff test to improve the measurement and reduce variability with pves.isv, therefore giving a more reproducible test. By improving the penile cuff test, the investigators can then go on to assess how our non-invasive measurements correlate with urodynamically derived indices of contractility, and use data from this pilot to help construct methodology of future cuff research. The current hypotheses are that; 1) accuracy of the cuff interruption pressure (pcuff.int) can be improved by modification of penile cuff test factors, 2) the number of valid inflations obtained per patient will increase with the modifications, and 3) that this non-invasive measure of contractility will correlate with pre-existing invasive indices.

The research protocol also gives the opportunity to explore correlation between commonly used symptom scores, and accuracy in the assessment of ultrasound residual urine volume measurement.

The primary objectives are therefore:

* To modify procedural steps of the penile cuff test that may reduce the previously observed variability and perform a pilot study to assess a reduction in variance
* To identify behaviour of the urethra during penile cuff inflation, by performing x-ray screening during the penile cuff test, and assess whether this is another source of inaccuracy
* To test the basic assumption of the penile cuff test that the bladder neck remains open during flow interruption

Secondary objectives of the study include the following:

* To compare non-invasive measurements from the penile cuff test against invasive indices of contractility
* To compare 2 different symptom scores for men with voiding lower urinary tract symptoms (LUTS)
* To assess accuracy and inter-observer variability of ultrasound residual measurement against a known volume.

ELIGIBILITY:
Inclusion Criteria:

* Male aged 18 years old or over
* Referred for video urodynamics within our department
* Predominant voiding LUTS as assessed by IPSS at screening. [The total IPSS score is out of 35, with up to 15 points for storage symptoms and 20 for voiding symptoms. If voiding symptoms as a percentage of total score is higher than storage symptoms they will be included in the study].
* Capacity to understand study procedures and give informed consent
* At least 2 voided volumes on frequency volume chart (FVC) of 250 mL

Exclusion Criteria:

* Female patients
* Long term catheterisation
* Predominant storage LUTS on IPSS at screening
* Fewer than 2 voids on FVC > 250 mL
* Known pre-existing neurological cause for symptoms
* Active urinary tract infection (UTI)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-08-28 (Actual); Primary Completion 2019-03 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Difference between invasive and non-invasive measurements | During the procedure
  Comparison of the pressure required to interrupt urine flow (pcuff.int) and simultaneously measured isovolumetric bladder pressure (pves.isv).

SECONDARY OUTCOMES:
Change in variance | During the procedure
  Comparison of results from this pilot study with analysis of past cohort to see if variances within the two populations are different (F test)
Assessment of bladder contractility - BCI | During the procedure
  Invasive assessment of contractility using the bladder contractility index (BCI). (it will also be analysed for correlation with pcuff.int)
Assessment of bladder contractility - Watt's Factor | During the procedure
  Invasive assessment of contractility using Watt's Factor (it will also be analysed for correlation with pcuff.int)
Quality of Life Assessment - ICIQ-MLUTS | During the procedure
  International Consultation on Incontinence Modular Questionnaire for male LUTS (ICIQ-MLUTS) will be completed by the participant. This is a modular symptom and quality of life questionnaire, in which the participant scores the frequency of a symptom from 0-4, and completes a 0-10 bother score (10 =worst) for each symptom. There are 20 questions in total. ( and analysed for correlation with outcome 6)
Quality of Life Assessment - IPSS | During the procedure
  International prostate symptoms score (IPSS) will be completed by the participant. Total score range 0-35 - generated from the sum of 7 questions related to urinary symptoms - all scored from 0-5 on degree of frequency. It will also be analysed for correlation with outcome 5)
Accuracy of ultrasound residual urine volume | During the procedure
  catheterized post void residual volume will be used as a gold standard to compare ultrasound residual measurements from two clinicians

CONTACTS AND LOCATIONS:
Overall Officials: Helen C Morton, MBBS, Principal Investigator — Newcastle upon Tyne Hospitals NHS Foundation Trust; Chris K Harding, MBBChir, MD, Study Director — Newcastle upon Tyne Hospitals NHS Foundation Trust; Alison Bray, PhD, Study Director — Newcastle upon Tyne Hospitals NHS Foundation Trust; James Blake, PhD, Study Director — Newcastle upon Tyne Hospitals NHS Foundation Trust
Locations (1):
- Freeman Hospital, Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle, Tyne and Wear, United Kingdom

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-05-15): https://cdn.clinicaltrials.gov/large-docs/15/NCT03603015/Prot_SAP_000.pdf
  • Informed Consent Form (2018-04-24): https://cdn.clinicaltrials.gov/large-docs/15/NCT03603015/ICF_001.pdf